CLINICAL TRIAL: NCT03228095
Title: Volatile Organic Compounds in Breath and Headspace Analysis - Diagnostic and Monitoring Markers for Diseases
Brief Title: Volatiles in Breath and Headspace Analysis - Diagnostic Markers
Acronym: Volatolome
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: University of Latvia (Other)
Collaborators: Technion, Israel Institute of Technology (Other); Riga East University Hospital (Unknown); JLM Innovation GmbH (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2017/20329
Record Dates: First submitted 2017-07-21; First posted 2017-07-24 (Actual); Last update posted 2018-08-21 (Actual); Status verified 2018-08

CONDITIONS: Tuberculosis; Gastric Cancer; Peptic Ulcer; Atrophic Gastritis; Intestinal Metaplasia; Gastric Dysplasia; Colorectal Cancer; Colorectal Polyp; Colorectal Adenoma; Pancreatic Cancer; Pancreatitis, Chronic; Liver Cancer; Liver Cirrhosis; Flu, Human; Other Infectious Diseases; Inflammatory Bowel Diseases
Keywords: Volatile Organic Compounds; Tuberculosis; Nano-sensors; Electronic nose; Digestive cancers
MeSH Terms: conditions — Tuberculosis; Stomach Neoplasms; Peptic Ulcer; Gastritis, Atrophic; Colorectal Neoplasms; Pancreatic Neoplasms; Pancreatitis, Chronic; Liver Neoplasms; Liver Cirrhosis; Influenza, Human; Inflammatory Bowel Diseases; Gastrointestinal Neoplasms | interventions — Gastroscopy; Biopsy; Colonoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Surgery and biopsy material as well as blood samples will contain himan DNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (17):
- Active Tuberculosis: Participants with Active Tuberculosis Disease Intervention: Diagnostic Test: VOC detection in breath and in skin headspace Procedure/Surgery: Whole blood/ Plasma / serum sampling Intervention: Diagnostic Test: Breath sampling Intervention: Headspace analysis for biological material
  Interventions: Diagnostic Test: VOC detection in breath and in skin headspace; Diagnostic Test: Breath sampling; Procedure: Whole blood/ Plasma / serum sampling; Diagnostic Test: Headspace analysis for biological material
- Group of Control (Tuberculosis): Participants Without Active Tuberculosis Disease Intervention: Diagnostic Test: VOC detection in breath and in skin headspace Procedure/Surgery: Whole blood/ Plasma / serum sampling Intervention: Diagnostic Test: Breath sampling Intervention: Headspace analysis for biological material
  Interventions: Diagnostic Test: VOC detection in breath and in skin headspace; Diagnostic Test: Breath sampling; Procedure: Whole blood/ Plasma / serum sampling; Diagnostic Test: Headspace analysis for biological material
- Gastric cancer: Patients with histologically confirmed gastric cancer Intervention: Diagnostic Test: Breath sampling Intervention: Procedure/Surgery: Upper endoscopy with biopsies Intervention: Procedure/Surgery: Whole blood/ Plasma / serum sampling Intervention: Diagnostic Test: Feacal sampling Intervention: Headspace analysis for biological material Intervention: Procedure/Surgery: Histological examination of surgical speciment
  Interventions: Diagnostic Test: Breath sampling; Procedure: Upper endoscopy with biopsies; Procedure: Whole blood/ Plasma / serum sampling; Diagnostic Test: Faecal sampling; Procedure: Histological examination of surgical specimen; Diagnostic Test: Headspace analysis for biological material
- Gastric dysplasia: Patients without gastric adenocarcinoma but with histologically confirmed dysplasia (either high- or low-grade) of the stomach Intervention: Diagnostic Test: Breath sampling Intervention: Procedure/Surgery: Upper endoscopy with biopsies Intervention: Procedure/Surgery: Whole blood/ Plasma / serum sampling Intervention: Headspace analysis for biological material Intervention: Diagnostic Test: Fecal sampling Intervention: Procedure/Surgery: Histological examination of surgical specimen
  Interventions: Diagnostic Test: Breath sampling; Procedure: Upper endoscopy with biopsies; Procedure: Whole blood/ Plasma / serum sampling; Diagnostic Test: Faecal sampling; Procedure: Histological examination of surgical specimen; Diagnostic Test: Headspace analysis for biological material
- High-risk gastric lesions: Patients graded Stage III-IV according to OLGIM (Operative Link of Gastric Intestinal Metaplasia Assessment) staging system, Stage III-IV according to OLGA (Operative Link for Gastric Atrophy Assessment), and those with incomplete type of intestinal metaplasia, but excluding those with dysplasia Intervention: Diagnostic Test: Breath sampling Intervention: Procedure/Surgery: Upper endoscopy with biopsies Intervention: Procedure/Surgery: Whole blood/ Plasma / serum sampling Intervention: Diagnostic Test: Fecal sampling Intervention: Procedure/Surgery: Histological examination of surgical specimen Intervention: Headspace analysis for biological material
  Interventions: Diagnostic Test: Breath sampling; Procedure: Upper endoscopy with biopsies; Procedure: Whole blood/ Plasma / serum sampling; Diagnostic Test: Faecal sampling; Procedure: Histological examination of surgical specimen; Diagnostic Test: Headspace analysis for biological material
- Normal and low-risk gastric lesions: Staged 0-III according to OLGIM. Dysplasia should be excluded Intervention: Diagnostic Test: Breath sampling Intervention: Procedure/Surgery: Upper endoscopy with biopsies Intervention: Procedure/Surgery: Whole blood/ Plasma / serum sampling Intervention: Diagnostic Test: Fecal sampling Intervention: Headspace analysis for biological material
  Interventions: Diagnostic Test: Breath sampling; Procedure: Upper endoscopy with biopsies; Procedure: Whole blood/ Plasma / serum sampling; Diagnostic Test: Faecal sampling; Diagnostic Test: Headspace analysis for biological material
- Colorectal cancer: Patients with histologically confirmed colorectal cancer (adenocarcinoma) Intervention: Diagnostic Test: Breath sampling Intervention: Procedure/Surgery: Colonoscopy with biopsies Intervention: Procedure/Surgery: Whole blood/ Plasma / serum sampling Intervention: Diagnostic Test: Fecal sampling Intervention: Headspace analysis for biological material Intervention: Procedure/Surgery: Histological examination of surgical specimen
  Interventions: Diagnostic Test: Breath sampling; Procedure: Colonoscopy with biopsies; Procedure: Whole blood/ Plasma / serum sampling; Diagnostic Test: Faecal sampling; Procedure: Histological examination of surgical specimen; Diagnostic Test: Headspace analysis for biological material
- Colorectal high-risk lesions: Patients without colorectal adenocarcinoma, but carrying high-risk adenomatous polyps being described by one of the following: 1) size≥1 cm; 2) high-grade dysplasia; 3) villous component. Prior to removal of the lesions Intervention: Diagnostic Test: Breath sampling Intervention: Procedure/Surgery: Colonoscopy with biopsies Intervention: Headspace analysis for biological material Intervention: Procedure/Surgery: Whole blood/ Plasma / serum sampling Intervention: Diagnostic Test: Fecal sampling Intervention: Procedure/Surgery: Histological examination of surgical specimen
  Interventions: Diagnostic Test: Breath sampling; Procedure: Colonoscopy with biopsies; Procedure: Whole blood/ Plasma / serum sampling; Diagnostic Test: Faecal sampling; Procedure: Histological examination of surgical specimen; Diagnostic Test: Headspace analysis for biological material
- Colorectal low-risk adenoma: Patients without colorectal adenocarcinoma and without colorectal high-risk lesions Intervention: Diagnostic Test: Breath sampling Intervention: Procedure/Surgery: Colonoscopy with biopsies Intervention: Procedure/Surgery: Whole blood/ Plasma / serum sampling Intervention: Diagnostic Test: Fecal sampling Intervention: Headspace analysis for biological material
  Interventions: Diagnostic Test: Breath sampling; Procedure: Colonoscopy with biopsies; Procedure: Whole blood/ Plasma / serum sampling; Diagnostic Test: Faecal sampling; Procedure: Histological examination of surgical specimen; Diagnostic Test: Headspace analysis for biological material
- Group of control (colorectal): Patients having undergone colonoscopy without an evidence for colorectal lesions Intervention: Diagnostic Test: Breath sampling Intervention: Procedure/Surgery: Colonoscopy with biopsies Intervention: Procedure/Surgery: Whole blood/ Plasma / serum sampling Intervention: Diagnostic Test: Fecal sampling Intervention: Headspace analysis for biological material Intervention: Procedure/Surgery: Histological examination of surgical specimen
  Interventions: Diagnostic Test: Breath sampling; Procedure: Colonoscopy with biopsies; Procedure: Whole blood/ Plasma / serum sampling; Diagnostic Test: Faecal sampling; Diagnostic Test: Headspace analysis for biological material
- Average risk general population: Average risk population of both genders aged 40-64 at the time of inclusion lacking alarm symptoms for gastrointestinal cancer Intervention: Diagnostic Test: Breath sampling Intervention: Procedure/Surgery: Whole blood/ Plasma / serum sampling Intervention: Diagnostic Test: Fecal sampling Intervention: Headspace analysis for biological material
  Interventions: Diagnostic Test: Breath sampling; Procedure: Whole blood/ Plasma / serum sampling; Diagnostic Test: Faecal sampling; Diagnostic Test: Headspace analysis for biological material
- Pancreatic cancer: Patients with histologically confirmed pancreatic cancer Intervention: Diagnostic Test: Breath sampling Intervention: Procedure/Surgery: Whole blood/ Plasma / serum sampling Intervention: Headspace analysis for biological material
  Interventions: Diagnostic Test: Breath sampling; Procedure: Whole blood/ Plasma / serum sampling; Procedure: Histological examination of surgical specimen; Diagnostic Test: Headspace analysis for biological material
- Chronic pancreatitis: Patients with clinically and/or histologically and/or radiologically confirmed chronic pancreatitis Intervention: Diagnostic Test: Breath sampling Intervention: Procedure/Surgery: Whole blood/ Plasma / serum sampling Intervention: Headspace analysis for biological material
  Interventions: Diagnostic Test: Breath sampling; Procedure: Whole blood/ Plasma / serum sampling; Diagnostic Test: Headspace analysis for biological material
- Liver cancer: Patients with histologically confirmed primary liver cancer Intervention: Diagnostic Test: Breath sampling Intervention: Procedure/Surgery: Whole blood/ Plasma / serum sampling Intervention: Headspace analysis for biological material
  Interventions: Diagnostic Test: Breath sampling; Procedure: Whole blood/ Plasma / serum sampling; Procedure: Histological examination of surgical specimen; Diagnostic Test: Headspace analysis for biological material
- Chronic liver disease: Patients with histologically confirmed liver cirrhosis of viral or other ethiology Intervention: Diagnostic Test: Breath sampling Intervention: Procedure/Surgery: Whole blood/ Plasma / serum sampling Intervention: Headspace analysis for biological material
  Interventions: Diagnostic Test: Breath sampling; Procedure: Whole blood/ Plasma / serum sampling; Diagnostic Test: Headspace analysis for biological material
- Upper respiratory tract acute infections: Patients with serologically confirmed infectious disease or individuals of high risk (e.g. population in season of flu epidemy). This group does not include tuberculosis Intervention: Diagnostic Test: Breath sampling Intervention: Procedure/Surgery: Whole blood/ Plasma / serum sampling Intervention: Headspace analysis for biological material
  Interventions: Diagnostic Test: Breath sampling; Procedure: Whole blood/ Plasma / serum sampling; Diagnostic Test: Headspace analysis for biological material
- Oncological diseases of other locations: Patients with histologically confirmed oncological diseases, excluding gastric, colorectal, pancreatic and primary liver cancer Intervention: Diagnostic Test: Breath sampling Intervention: Procedure/Surgery: Whole blood/ Plasma / serum sampling Intervention: Headspace analysis for biological material
  Interventions: Diagnostic Test: Breath sampling; Procedure: Whole blood/ Plasma / serum sampling; Procedure: Histological examination of surgical specimen; Diagnostic Test: Headspace analysis for biological material

INTERVENTIONS:
Diagnostic Test: VOC detection in breath and in skin headspace — VOC will be detected in breath with off-line and on-line testing and in skin headspace with off-line testing
  Groups: Active Tuberculosis; Group of Control (Tuberculosis)
Diagnostic Test: Breath sampling — Breath sampling for VOCs detections will be carried out using nano-sensor based devices (electronic nose)
Procedure: Upper endoscopy with biopsies — Upper endoscopy with proper biopsy work-up will be used for identification and stratification of gastric lesions as well as acquisition of biopsies for microbiota testing
  Groups: Gastric cancer; Gastric dysplasia; High-risk gastric lesions; Normal and low-risk gastric lesions
Procedure: Colonoscopy with biopsies — Colonoscopy with proper biopsy or polypectomy material work-up will be used for identification and stratification of colorectal lesions as well as acquisition of biopsies for microbiota testing
  Groups: Colorectal cancer; Colorectal high-risk lesions; Colorectal low-risk adenoma; Group of control (colorectal)
Procedure: Whole blood/ Plasma / serum sampling — Whole blood/Plasma/serum sampling will be used to obtain information for group stratification
Diagnostic Test: Faecal sampling — Facal samples will be obtained for faecal occult blood testing as well as microbiota analysis
  Groups: Average risk general population; Colorectal cancer; Colorectal high-risk lesions; Colorectal low-risk adenoma; Gastric cancer; Gastric dysplasia; Group of control (colorectal); High-risk gastric lesions; Normal and low-risk gastric lesions
Procedure: Histological examination of surgical specimen — Routine histological exam for patients undergoing curative or palliative surgery. Indication for surgery are set based on underlying condition. Study does not interfere with decision making for surgical treatment
  Groups: Colorectal cancer; Colorectal high-risk lesions; Colorectal low-risk adenoma; Gastric cancer; Gastric dysplasia; High-risk gastric lesions; Liver cancer; Oncological diseases of other locations; Pancreatic cancer
Diagnostic Test: Headspace analysis for biological material — VOC analysis from headspace of surgical specimen, biopsy materials, blood/plasma, microbiota etc.

SUMMARY:
Detection of Volatile Organic Compounds (VOC) directly from tissue by headspace analysis (skin, surgery material, other tissue) and exhaled breath is feasible using affordable user-friendly novel nano-chemo sensors that can accurately be used for screening and monitoring purpose

DETAILED DESCRIPTION:
Study propose to explore a novel approach for the diagnosis and monitoring of diseases. The approach is based on the detection of volatile organic compounds (VOCs) that are emitted from the cells and detected directly from tissue, such as skin, surgery material, blood as well as from exhaled breath.

In the literature there are several reports on VOCs which can be detected by Gas Chromatography - Mass Spectrometry (GC-MS) means directly from: (i) the headspace of TB cells (i.e., the mixture of volatile biomarkers trapped above the TB cells in a sealed vessel); (ii) the exhaled breath or (iii) from urine. Excellent results in detection of the tuberculosis disease by using nanosensor array were shown by Nakhleh et al achieved 90% sensitivity, 93% specificity and 92% accuracy in discrimination between healthy and diseased patients using electronic nose devices with a single sensor. None of the reported studies identified the tentative recognition of the tuberculosis-related VOCs and quantified the concentration differences between samples from ill and healthy controls. Further investigation of the exhaled breath tuberculosis-related VOC by GC-MS means will improve the knowledge and simultaneously will help to improve the nanosensor array design.

Several studies have shown that disease-rated VOC patterns can be transmitted through the skin, and, therefore, skin can be used as a source for disease detection and identification. The principle of this detection approach is that disease-related changes are reflected in measurable changes in the skin through exchange via the blood. In addition, several studies have suggested that the VOC levels are elevated even in early stages of the disease, because they reflect a change in the human's body chemistry (as a result of the development of disease condition), rather than the amount of infected cells. Complementary studies have shown that VOCs can be emitted to the skin within minutes after they have emerged in the infected part of the human's body. What is particularly significant about this approach is that each type of (infectious) disease has its own unique pattern of VOCs, and, therefore, the presence of one (infectious) disease would not screen other disease types. Nevertheless, to the best of our knowledge, the detection of tuberculosis VOCs through skin has not been examined yet. Additionally, all studies targeting skin VOCs have been carried out by means of spectrometry and spectroscopy techniques. In few cases, electronic nose devices were used. These techniques are powerful tools for detecting VOCs. However, to date, the use of these techniques has been impeded by the need for moderately to highly expensive equipment's, the high levels of expertise required to operate such instruments, the speed required for sampling and analysis, and the need for preconcentration techniques. For VOC skin testing and breath testing of tuberculosis to become widely used in clinical practice, several advances in the knowledge of tuberculosis specific VOCs and sensor development need to occur. Nanoparticles containing flexible sensors, based on organic films, are more likely to become a clinical diagnostic tool, because they are significantly smaller, easier-to-use, and significantly less expensive.

In recent years comprehensive studies have shown excellent data for using VOCs from exhaled breath as tool for diagnosing gastric cancer. In one of the biggest studies carried out by Chinese and Latvian centers, malignancy could be identified with 89% sensitivity and 90% specificity after cross-validation, irrespective of important confounding factors in gastric patients such as tobacco or alcohol consumption and H. pylori infection. A breath test for GC staging could also be demonstrated by distinguishing stage I&II cancers from stage III&IV cancers with 89% sensitivity and 94% specificity. These studies used both - mass spectometry and nano-sensors technologies. Most recent study published in ASC Nano journal in January 2017 reported on more extended use of nanoarry sensors in breath analysis, blind experiments showed that 86% accuracy could be achieved with the artificially intelligent nanoarray, allowing both detection and discrimination between the different disease conditions examined (chronic kidney failure, idiopathic Parkinson's disease, atypical Parkinsonism , multiple sclerosis, Crohn's disease, ulcerative colitis, irritable bowel syndrome, pulmonary arterial hypertension, pre-eclampsia in pregnant women, head and neck cancer, lung cancer, colorectal cancer, bladder cancer, kidney cancer, prostate cancer, gastric cancer, and ovarian cancer. Analysis of the artificially intelligent nanoarray also showed that each disease has its own unique breathprint, and that the presence of one disease would not screen out others.

Therefore, this study is aimed to test VOCs detecting technologies as diagnostic and monitoring tools for digestive tract and infectious diseases.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent signed
* Individual with targeted disease/lesion (tuberculosis, gastric cancer, gastric dysplasia, high/ normal/ low risk gastric lesions, colorectal cancer, high-risk colorectal lesions, low-risk colorectal adenoma, pancreatic cancer, chronic pancreatitis, liver cancer, chronic liver disease, other infectious diseases, oncological diseases of other location)

Exclusion Criteria:

* Informed Consent not signed
* Other active cancer at the time of inclusion for particular study group

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients being referred for diagnostic testing and treatment Healthy individuals from general population
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2017-07-24 (Actual); Primary Completion 2019-12-20 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Specific VOC detected | 2 years
  Tuberculosis specific VOC detected in breath and in skin headspace
Performance of nanoarray sensor testing to detect target lesions and diseases | At the time of breath sampling
  Sensitivity, specificity, overall accuracy of nanoarray sensor testing for VOCs to detect the target lesions in the blinded analysis

SECONDARY OUTCOMES:
Specific VOC patterns for target disease or lesion and risk groups | At the time of breath sampling
  List of VOCs assayed by GC-MS with statistical difference between the study groups
VOC pattern changes following treatment | At baseline, 3 and/or 6 months after treatment (other time frame according to study group)
  VOC pattern changes after specific required treatment (medical eradication of bacteria/viruses, surgery/endoscopic removal for cancers or high risk lesion)
VOC pattern changes in relapse of disease for early recognition and treatment | At baseline, 3 and/or 6 months after treatment (other time frame according to study group)
  VOC pattern changes at the time of surveillance in case of relapse (malignant diseases).
Groups of gastrointestinal microbiota correlating to VOCs | At the time of sampling
  List of gastrointestinal microbiota groups (phylum/genus level) with positive correlation to particular VOCs

CONTACTS AND LOCATIONS:
Overall Officials: Mārcis Leja, PhD, MD, Study Director — University of Latvia; Lelde Lauka, MD, Principal Investigator — University of Latvia; Andra Cīrule, MD, Principal Investigator — Riga East University Hospital
Locations (1):
- University of Latvia, Riga, Latvia

REFERENCES:
- [Background] Nakhleh MK, Amal H, Jeries R, Broza YY, Aboud M, Gharra A, Ivgi H, Khatib S, Badarneh S, Har-Shai L, Glass-Marmor L, Lejbkowicz I, Miller A, Badarny S, Winer R, Finberg J, Cohen-Kaminsky S, Perros F, Montani D, Girerd B, Garcia G, Simonneau G, Nakhoul F, Baram S, Salim R, Hakim M, Gruber M, Ronen O, Marshak T, Doweck I, Nativ O, Bahouth Z, Shi DY, Zhang W, Hua QL, Pan YY, Tao L, Liu H, Karban A, Koifman E, Rainis T, Skapars R, Sivins A, Ancans G, Liepniece-Karele I, Kikuste I, Lasina I, Tolmanis I, Johnson D, Millstone SZ, Fulton J, Wells JW, Wilf LH, Humbert M, Leja M, Peled N, Haick H. Diagnosis and Classification of 17 Diseases from 1404 Subjects via Pattern Analysis of Exhaled Molecules. ACS Nano. 2017 Jan 24;11(1):112-125. doi: 10.1021/acsnano.6b04930. Epub 2016 Dec 21. PMID 28000444
- [Background] Xu ZQ, Broza YY, Ionsecu R, Tisch U, Ding L, Liu H, Song Q, Pan YY, Xiong FX, Gu KS, Sun GP, Chen ZD, Leja M, Haick H. A nanomaterial-based breath test for distinguishing gastric cancer from benign gastric conditions. Br J Cancer. 2013 Mar 5;108(4):941-50. doi: 10.1038/bjc.2013.44. PMID 23462808
- [Background] Amal H, Leja M, Broza YY, Tisch U, Funka K, Liepniece-Karele I, Skapars R, Xu ZQ, Liu H, Haick H. Geographical variation in the exhaled volatile organic compounds. J Breath Res. 2013 Dec;7(4):047102. doi: 10.1088/1752-7155/7/4/047102. Epub 2013 Nov 1. PMID 24184568